CLINICAL TRIAL: NCT04271670
Title: Effect of Warm Water Footbaths With Added Ginger or Mustard Powder on Psychosocial Parameters in Patients With an Oncological Disease: a Randomized Controlled Trial
Brief Title: Effect of Warm Water Footbaths With Added Ginger or Mustard Powder on Psychosocial Parameters in Patients With an Oncological Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SWI_03
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Oncologic Disorders
Keywords: Ginger; Mustard; Footbath; Warmth perception; Infrared thermography; Healthy volunteers

STUDY DESIGN:
Intervention Model Description: Each participant receives all three footbath interventions (warm water only=WA, with added ginger powder=GI, with added mustard powder=MU) in a randomized order stratified by gender. For this, participants are randomly allocated to one of six possible footbath sequences (a: MU-WA-GI, b: MU-GI-WA, c: WA-GI-MU, d: WA-MU-GI, e: GI-MU-WA, f: GI-WA-MU). For the main analysis, groups are pooled together with regard to the intervention received (WA vs. MU vs. GI) after checking for potential carry-over effects.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Warm water footbath with ginger powder (Experimental): Footbath with ginger powder with a maximum duration of 20 minutes.
  Interventions: Other: Ginger powder footbaths
- Warm water footbath with mustard powder (Experimental): Footbath with mustard powder with a maximum duration of 20 minutes.
  Interventions: Other: Mustard powder footbaths
- Warm water only footbath (Active Comparator): Warm water only footbath with a maximum duration of 20 minutes.
  Interventions: Other: Warm water only footbaths

INTERVENTIONS:
Other: Ginger powder footbaths — 20-minute footbath with 12 liters of 40°C warm water and an additive of 80g dried ginger powder (reaching up to mid-calf level)
  Arms: Warm water footbath with ginger powder
Other: Mustard powder footbaths — 20-minute footbath with 12 liters of 40° C warm water and an additive of 80g dried mustard powder (reaching up to mid-calf level)
  Arms: Warm water footbath with mustard powder
Other: Warm water only footbaths — 20-minute footbath with 12 liters of 40° C warm water without any additive (reaching up to mid-calf level)
  Arms: Warm water only footbath

SUMMARY:
A randomized, controlled, three-arm trial to investigate the effects of warm water footbaths with and without the addition of ginger or mustard powder on psychosocial parameters in patients with an oncological disease and in healthy controls.

DETAILED DESCRIPTION:
A randomized, controlled trial with cross-over design in which the subjects (23 patients with an oncological disease, 13 healthy controls) receive warm water footbaths with added ginger (experimental) or mustard powder (experimental) or without additives (active comparator). The wash-out period between two consecutive footbath interventions is at least one day. Outcome measures are assessed right before (t1), right after (t2) and 10 minutes following the footbath (t3). The main focus is on the change in subjective perception of warmth distribution between t1 and t3. Moreover, the objective skin temperature distribution and psychosocial scores are assessed. The primary outcome measure is analyzed with a linear mixed effects model (after checking for carry-over effects). Secondary outcome measures are described descriptively.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 18 and 65 years
* Oncological disorder with at least one chemotherapy or radiation in the treatment history
* Current inpatient treatment in the oncology ward of the Filderklinik (Filderstadt, Germany) with a minimum stay of 4 days

Exclusion Criteria:

* Infectious disease (with more than 38 °C core body temperature)
* Skin lesion on the lower legs or feet
* Hypersensitivity to mustard or ginger products
* Cardiac arrhythmia
* Pregnancy
* Insufficient knowledge of the German language
* Bedriddenness
* Poor general condition (according to the assessment of the attending physicians)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Change in subjective feeling of warmth at the feet as assessed by the "Herdecke Warmth Perception Questionnaire" from t1 to t3 | Immediately before the footbath (t1) and 10 minutes following the footbath (t3)
  Self-reported feeling of warmth at the feet, measured with the "Herdecke Warmth Perception Questionnaire", score between 0=cold and 4=hot

SECONDARY OUTCOMES:
Change in subjective feeling of warmth at the feet as assessed by the "Herdecke Warmth Perception Questionnaire" from t1 to t2 | Immediately before the footbath (t1) and immediately after the footbath (t2)
  Self-reported feeling of warmth at the feet, measured with the "Herdecke Warmth Perception Questionnaire", score between 0=cold and 4=hot
Change in subjective feeling of warmth in the face as assessed by the "Herdecke Warmth Perception Questionnaire" from t1 to t3 | Immediately before the footbath (t1) and 10 minutes following the footbath (t3)
  Self-reported feeling of warmth in the face, measured with the "Herdecke Warmth Perception Questionnaire", score between 0=cold and 4=hot
Change in subjective feeling of warmth in the face as assessed by the "Herdecke Warmth Perception Questionnaire" from t1 to t2 | Immediately before the footbath (t1) and immediately after the footbath (t2)
  Self-reported feeling of warmth in the face, measured with the "Herdecke Warmth Perception Questionnaire", score between 0=cold and 4=hot
Change in subjective feeling of warmth at the hands as assessed by the "Herdecke Warmth Perception Questionnaire" from t1 to t3 | Immediately before the footbath (t1) and 10 minutes following the footbath (t3)
  Self-reported feeling of warmth at the hands, measured with the "Herdecke Warmth Perception Questionnaire", score between 0=cold and 4=hot
Change in subjective feeling of warmth at the hands as assessed by the "Herdecke Warmth Perception Questionnaire" from t1 to t2 | Immediately before the footbath (t1) and immediately after the footbath (t2)
  Self-reported feeling of warmth at the hands, measured with the "Herdecke Warmth Perception Questionnaire", score between 0=cold and 4=hot
Change in subjective feeling of overall warmth as assessed by the "Herdecke Warmth Perception Questionnaire" from t1 to t3 | Immediately before the footbath (t1) and 10 minutes following the footbath (t3)
  Self-reported feeling of overall warmth, measured with the "Herdecke Warmth Perception Questionnaire", score between 0=cold and 4=hot
Change in subjective feeling of overall warmth as assessed by the "Herdecke Warmth Perception Questionnaire" from t1 to t2 | Immediately before the footbath (t1) and immediately after the footbath (t2)
  Self-reported feeling of overall warmth, measured with the "Herdecke Warmth Perception Questionnaire", score between 0=cold and 4=hot
Warmth perception and skin stimulus at the feet during the footbath | Up to 20 minutes
  Self-reported perception of warmth and skin stimulus during the footbath, assessed with a dynamic warmth and skin stimulus visual analog scale (VAS), applied once per minute (0 = cold/no stimulus; 10 = very hot/very strong stimulus)
Change in well-being from t1 to t2 | Immediately before (t1) and immediately after the footbath (t2)
  Self-reported well-being, assessed with the "Basler Befindlichkeits-Skala" (Basel Mood Questionnaire, BBS; 16 items; 7-point rating scale; higher values
Change in well-being from t1 to t3 | Immediately before (t1) and ten minutes following the footbath (t3)
  Self-reported well-being, assessed with the "Basler Befindlichkeits-Skala" (Basel Mood Questionnaire, BBS; 16 items; 7-point rating scale; higher values represent a better outcome)
Change in skin temperature at the feet from t1 to t3 | Immediately before (t1) and ten minutes following the footbath (t3)
  Skin temperature (in °C) at both feet, measured with a high-definition infrared camera (FLIR-Systems, type SC660)
Change in skin temperature at the feet from t1 to t2 | Immediately before the footbath (t1) and immediately after the footbath (t2)
  Skin temperature (in °C) at both feet, measured with a high-definition infrared camera (FLIR-Systems, type SC660)
Change in skin temperature at the hands from t1 to t3 | Immediately before (t1) and ten minutes following the footbath (t3)
  Skin temperature (in °C) at both hands, measured with a high-definition infrared camera (FLIR-Systems, type SC660)
Change in skin temperature at the hands from t1 to t2 | Immediately before the footbath (t1) and immediately after the footbath (t2)
  Skin temperature (in °C) at both hands, measured with a high-definition infrared camera (FLIR-Systems, type SC660)
Change in skin temperature in the face from t1 to t3 | Immediately before (t1) and ten minutes following the footbath (t3)
  Skin temperature (in °C) in the face, measured with a high-definition infrared camera (FLIR-Systems, type SC660)
Change in skin temperature in the face from t1 to t2 | Immediately before the footbath (t1) and immediately after the footbath (t2)
  Skin temperature (in °C) in the face, measured with a high-definition infrared camera (FLIR-Systems, type SC660)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, MD, Study Director — ARCIM Institute
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.